CLINICAL TRIAL: NCT03403725
Title: Open-Label, Multicenter, Phase I Dose Escalation Study of MEN1309, a CD205 Antibody-Drug Conjugate,in Patients With CD205-Positive Metastatic Solid Tumors and Non-Hodgkin Lymphoma
Brief Title: MEN1309 I.v. Infusion in Pts With CD205-positive Metastatic Solid Tumors and Relapsed or Refractory NHL Ph I Study
Acronym: CD205SHUTTLE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated after achievement of MTD, without progressing to cohort expansion for Company decision.
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEN1309-01
Record Dates: First submitted 2018-01-04; First posted 2018-01-19 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Solid Tumors; Relapsed/Refractory Non-Hodgkin Lymphoma
Keywords: Solid Tumors; Non-Hodgkin Lymphoma; NHL; MEN1309; CD205; Relapsed; Refractory; R-R NHL; ADC; Antibody-Drug Coniugate; Metastatic Tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Cohort1 0.05mg/kg STEP 1 Solid Tumors Cohort2 0.10mg/kg STEP 1 Solid Tumors Cohort3 0.20mg/kg STEP 1 Solid Tumors Cohort4 0.40mg/kg STEP 1 Solid Tumors Cohort5 0.80mg/kg STEP 1 Solid Tumors Cohort6 1.60mg/kg STEP 1 Solid Tumors Cohort7 2.40mg/kg STEP 1 Solid Tumors Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF Cohort5 0.80mg/kg STEP 2 NHL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEN1309 (Step 1-Solid Tumors)/(Step 2-NHL) (Experimental): Step1: Accelerated Titration Design with 1 single pt per cohort and double dose level per cohort until grade ≥ 2 drug related toxicity. Then, study reverts to 3+3 design. Any cohort in which 1 pt experiences a DLT (along ATD or 3+3) will be expanded up to 6 pts.
  Step2: MTD defined in Step 1, 3 MEN1309 dose levels will be tested (MTD-2, MTD-1, and MTD), with 6 pts per each dose level. A further MTD-3 level will be explored if 2 DLTs occur at the MTD-2 dose level.
  Interventions: Drug: MEN1309

INTERVENTIONS:
Drug: MEN1309 — MEN1309 solution for intravenous infusion once every 3 weeks

SUMMARY:
The purpose of this clinical trial is to identify the highest dose of MEN1309 drug with acceptable safety profile and that can be used in patients affected by CD205-positive solid tumors and Non-Hodgkin Lymphoma

DETAILED DESCRIPTION:
This clinical trial will investigate the safety and activity of MEN1309 in patients with CD205-positive metastatic solid tumors and Non-Hodgkin Lymphoma who have tried other types of treatment for cancer without adequate response (or the cancer came back). CD205 is a protein present in certain types of cancer.

This is a Phase I study, which means that it is designed to look at several dose levels of a study drug in small groups of patients to find the dose that is well-tolerated and suitable to be administered in subsequent clinical trials in patients. The clinical trial is also looking at the effectiveness of the study drug. This is the first time the study drug will be given in humans.

The clinical trial consists of two sequential parts:

* Part 1 involves patients with CD205-positive metastatic solid tumors and the main purpose of this part of the clinical trial is to determine the highest dose of the study drug that can be used safely in these type of cancers.
* Part 2 involves patients with CD205-positive Non-Hodgkin Lymphoma and will test doses of MEN1309 which have demonstrated to be adequately tolerated in patients with solid tumors.

Patients participating to the clinical trial will take the study drug as intravenous infusion once every 3 weeks. The clinical trial includes four periods: a pre-screening period (to check if tumor is positive for CD205), a screening period (to check whether the participation to the clinical trial is right for patient), a treatment period (when patient receives the study drug), and a follow-up period (to check the health status of the patient after stopping study treatment).

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female patients aged ≥ 18 years.
2. Patients with:

   * confirmed diagnosis of advanced or metastatic solid tumor and diagnosis of multiple relapsed or refractory NHL;
   * progressive after last treatment received;
   * availability of archived tumor material, either as a block or slides;
   * measurable or evaluable disease by Response Evaluation Criteria in solid tumors guideline (RECIST v1.1) and by Cheson Criteria (The Lugano Classification, 2014) in NHL.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
4. Neutrophil count ≥ 1,500/µL; platelets ≥ 100,000/µL; haemoglobin ≥ 9 g/dL.
5. Adequate renal and hepatic laboratory assessments.
6. Life expectancy of at least 2 months.
7. Woman of childbearing potential (WOCBP) who agrees to use highly effective contraception (see Appendix I).

Main Exclusion Criteria:

1. Central nervous system involvement (excluding treated stable cerebral metastasis, not requiring therapy to control symptoms in the last 60 days).
2. Pregnant or breastfeeding women.
3. Life-threatening illnesses other than solid tumors and NHL, uncontrolled medical conditions or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety, or put the study outcomes at risk.
4. Less than 2 previous cancer treatments, including high dose chemotherapy and ASCT, for NHL unless patient refuses standard therapy and/or is not eligible for ASCT.
5. Have significant, uncontrolled, or active cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero Head, Medical Oncology Department, MD PhD, Study Chair — Vall d' Hebron Institute of Oncology (VHIO) P. Vall d'Hebron 119-129 08035 Barcelona, Spain
Locations (7):
- CHU Sart Tilman, Liège, Belgium
- Italy (2):
  - Centro Riferimento Oncologico, Aviano
  - IRCCS Ospedale San Raffaele, Milan
- Spain (3):
  - Vall d'Hebron Barcelona Hospital, Barcelona
  - START Madrid. Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
- NCCC Clinical Trials Pharmacy, Northern Centre for Cancer Care, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to perform this study in 7 sites across 4 European countries: Spain, Italy, Belgium, and UK. Patients were only recruited in 5 sites (3 ES, 1 IT1, 1 BE) prior to the study being stopped. The study started in date 28 August 2017 (FPI) to 19 November 2019 (LPLV). Study Termination letter was sent to authorities on 08 January 2020.
Pre-assignment Details: Male or female patients aged ≥ 18 years. For Step 1 of the study, patients with diagnosis of advanced or metastatic solid tumor. For Step 2, patients with histologically confirmed diagnosis of relapsed or refractory NHL. In both Steps the tumor need to have a positivity (≥ 1+ IHC staining) for CD205.
Groups:
- Cohort1 0.05mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved a dose of 0.05 mg/Kg of MEN1309.
- Cohort2 0.10mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved a dose of 0.10 mg/Kg of MEN1309.
- Cohort3 0.20mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved a dose of 0.20 mg/Kg of MEN1309.
- Cohort4 0.40mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved a dose of 0.40 mg/Kg of MEN1309.
- Cohort5 0.80mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved a dose of 0.80 mg/Kg of MEN1309.
- Cohort6 1.60mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved a dose of 1.60 mg/Kg of MEN1309.
- Cohort7 2.40mg/kg STEP 1 Solid Tumors; Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF: Patients with CD205-positive advanced solid tumors, who recieved a dose of 2.40 mg/Kg of MEN1309.
- Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF: Patients with CD205-positive advanced solid tumors, who recieved a dose of 3.36 mg/Kg of MEN1309.
- Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF: Patients with CD205-positive advanced solid tumors, who recieved a dose of 2.00 mg/Kg of MEN1309.
- Cohort5 0.80mg/kg STEP 2 NHL: Patients with CD205-positive multiple relapsed or refractory Non Hodking Lymphoma, who recieved a dose of 0.80 mg/Kg of MEN1309.
Period: Overall Study
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Started | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort1 0.05mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved 0.05mg/kg of MEN1309.
- Cohort2 0.10mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved 0.10mg/kg of MEN1309.
- Cohort3 0.20mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved 0.20mg/kg of MEN1309.
- Cohort4 0.40mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved 0.40mg/kg of MEN1309.
- Cohort5 0.80mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved 0.80mg/kg of MEN1309.
- Cohort6 1.60mg/kg STEP 1 Solid Tumors: Patients with CD205-positive advanced solid tumors, who recieved 1.60mg/kg of MEN1309.
- Cohort7 2.40mg/kg STEP 1 Solid Tumors; Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF: Patients with CD205-positive advanced solid tumors, who recieved 2.40mg/kg of MEN1309.
- Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF: Patients with CD205-positive advanced solid tumors, who recieved 3.36mg/kg of MEN1309.
- Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF: Patients with CD205-positive advanced solid tumors, who recieved 2.00mg/kg of MEN1309.
- Cohort5 0.80mg/kg STEP 2 NHL: Patients with CD205-positive multiple relapsed or refractory Non Hodking Lymphoma, who recieved 0.80mg/kg of MEN1309.
- Total: Total of all reporting groups
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 1 | 4 | 3 | 2 | 2 | 2 | 0 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 2 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 0 | 3 | 6 | 3 | 1 | 2 | 0 | 19
  Male | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 2 | 1 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 2 | 3 | 1 | 26
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 5
  Italy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Spain | 1 | 1 | 1 | 1 | 0 | 5 | 5 | 2 | 2 | 3 | 1 | 0
Weight [Mean (Standard Deviation); unit: Kg] | 66.10 (0) | 56.80 (0) | 60.60 (0) | 62.50 (0) | 53.50 (0) | 64.27 (17.382) | 67.30 (15.725) | 61.17 (8.520) | 76.57 (15.584) | 64.55 (8.805) | 109.4 (0) | 66.68 (12.886)

OUTCOME MEASURES:

1. Primary Outcome: Maximum-Tolerated Dose (MTD)
Description: Defined as the highest dose level at which no more than 1 of 6 patients experiences a DLT during the DLT assessment window.
Time Frame: 21-day period after the first dose
Population: MTD was evaluated only in the STEP 1 since in STEP 2 only one patient was treated.
Measure: Number; unit: mg/Kg
Groups:
- All Doses STEP 1-Solid Tumors: All Patients with CD205-positive advanced solid tumors inlcuded in STEP1.
Arm/Group | All Doses STEP 1-Solid Tumors
Number analyzed (Participants) | 27
mg/Kg | 1.6

2. Primary Outcome: Dose-Limiting Toxicity (DLT)
Description: Adverse drug reactions (ADRs) that will be assessed during Cycle 1:
  * any grade ≥ 3 cardiac toxicity, new segmental wall-motion abnormalities, or cardiac troponin I or T elevation of grade 3 or higher;
  * any grade ≥ 3 elevations in total bilirubin, hepatic transaminases, or ALP levels; in patients with baseline grade 2 hepatic transaminase or ALP levels, an elevation to ≥ 10 x ULN is considered a DLT;
  * any grade 3 non-haematologic toxicity lasting > 7 days, (excluding diarrhea/nausea for which no adequate and optimal therapy has been implemented and alopecia);
  * any grade 3 vomiting lasting > 3 days despite adequate and optimal therapy;
  * any grade ≥ 4 non-haematologic toxicity;
  * any grade 4 thrombocytopenia or anemia;
  * any grade 4 neutropenia lasting > 7 days or febrile neutropenia;
  * any treatment delay of > 2 weeks because of delayed recovery from toxicity related to MEN1309 (except for alopecia).
Time Frame: 21-day period after the first dose
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
Dose Limiting Toxicities | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 0

3. Secondary Outcome: Overall Survival
Description: Timeframe between the first study drug administration and death from any cause.
Time Frame: Through study completion, from "August 28, 2017" to "January 8, 2020" (2 years and 4 months)
Population: For Cohorts reported as 0 analyzed the patients were censored (Event Date Not available)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 3 | 0
Days |  | 379 (0) | 700 (0) |  | 74 (0) | 154 (0) | 297.75 (208.73) |  |  | 90.33 (12.66) |

4. Secondary Outcome: Progression Free Survival
Description: The Number of days between the first study administration to the date of first documented disease progression.
Time Frame: Through study completion, from "August 28, 2017" to "January 8, 2020" (2 years and 4 months)
Population: For Cohorts reported as 0 analyzed the patients were censored (Event Date Not available)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 2 | 3 | 0
Days |  |  | 41 (0) |  | 38 (0) | 36.5 (0.71) | 155.5 (190.51) |  | 100.5 (28.99) | 37 (1.73) |

5. Secondary Outcome: Preliminary Tumor Activity (RR)
Description: Preliminary tumor activity (RR) Response Rate. RECIST v 1.1 assessment was performed using CT or MRI scan of the chest and abdomen (including adrenal glands). For the baseline assessment, CT or MRI scan were to be performed no more than 6 weeks (4+2 weeks) before the treatment start. Follow-up assessment were performed every other cycle starting from cycle 3 until the End of Study Visit.
Time Frame: From Day1Visit1 to End of the treatment (At Baseline no more than 6 weeks before treatment and then every cycle starting from cycle 3 until End of Study)
Population: Efficacy Population:All eligible patients who receive at least 2 complete treatment cycles and have at least 1 disease assessment are to be considered evaluable for efficacy.
  The percentage of patient is 0% since no patient had Complete response or partial response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Preliminary Antitumor Activity (DCR)
Description: Preliminary Antitumor Activity (DCR) Disease control Rate. RECIST v 1.1 assessment was performed using CT or MRI scan of the chest and abdomen (including adrenal glands). For the baseline assessment, CT or MRI scan were to be performed no more than 6 weeks (4+2 weeks) before the treatment start. Follow-up assessment were performed every other cycle starting from cycle 3 until the End of Study Visit.
Time Frame: as for outcome 5
Population: Efficacy Population:All eligible patients who receive at least 2 complete treatment cycles and have at least 1 disease assessment are to be considered evaluable for efficacy.
  Out of 11 evaluable patients, 11 patients had stable disease (SD), no complete response or partial response was observed.
Measure: Number; unit: N. of Stable Disease/N. of Pts
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 2 | 4
N. of Stable Disease/N. of Pts | 0 | 0 | 0 |  | 1 |  | 0.33 | 0.8 |  | 0 | 0.25

7. Secondary Outcome: Preliminary Antitumor Activity (DOR)
Description: Prliminary Antitumor Activity. Measure of the Duration of response. RECIST v 1.1 assessment was performed using CT or MRI scan of the chest and abdomen (including adrenal glands). For the baseline assessment, CT or MRI scan were to be performed no more than 6 weeks (4+2 weeks) before the treatment start. Follow-up assessment were performed every other cycle starting from cycle 3 until the End of Study Visit.
Time Frame: as for outcome 5
Population: Data Cannot be reported since it was not analyzed. No Patients had Complete response and Partial Response.
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: MEN1309 PK Parameter Cmax
Description: Cmax is the maximum drug concentration
Time Frame: Cycle 1
Measure: Mean (Standard Deviation); unit: microgram/mL
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
microgram/mL | 0.73 (0.19) | 0.87 (0.16) | 1.75 (0.09) | 3.16 (0) | 9.67 (2.03) | 31.87 (9.11) | 43.94 (11.25) | 64.97 (33.40) | 44.50 (15.79) | 33.52 (9.29) | 11.36 (0)

9. Secondary Outcome: MEN1309 PK Parameter Ctrough
Description: MEN1309 PK parameter Ctrough (Predose concentration)
Time Frame: Pre-infusion Cycle 2
Population: For Cohort 4 the treatment ended at Cycle 1 for the only subejct.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 6 | 6 | 3 | 3 | 4 | 1
ng/mL | 0 (0) | 0 (0) | 0 (0) |  | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

10. Secondary Outcome: MEN1309 Pharmacokinetic (PK) Parameter t1/2
Description: MEN1309 Pharmacokinetic (PK) parameter t1/2 (terminal serum half-life)
Time Frame: Cycle 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
hr | 2.66 (0) | 3.17 (0) | 2.38 (0) | 16.65 (0) | 93.90 (0) | 18.24 (6.49) | 16.89 (1.67) | 27.74 (2.36) | 15.36 (0.96) | 17.24 (1.24) | 15.08 (0)

11. Secondary Outcome: MEN1309 Pharmacokinetic (PK) Parameter AUC
Description: MEN1309 Pharmacokinetic (PK) parameter AUC (area under curve)
Time Frame: Cycle 1
Measure: Mean (Standard Deviation); unit: hr * microgram/mL
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
hr * microgram/mL | 3.94 (0) | 3.78 (0) | 6.16 (0) | 11.86 (0) | 57.49 (0) | 583.38 (213.45) | 1038.12 (257.12) | 2045.41 (1130.69) | 958.94 (417.06) | 689.33 (295.50) | 111.44 (0)

12. Secondary Outcome: MEN1309 (PK) Parameter CL
Description: Systemic clearance of MEN1309 Pharmacokinetic
Time Frame: Cycle 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
L/hr | 0.82 (0) | 1.46 (0) | 1.96 (0) | 2.06 (0) | 0.70 (0) | 0.20 (0.09) | 0.17 (0.08) | 0.13 (0.9) | 0.21 (0.07) | 0.22 (0.11) | 0.78 (0)

13. Secondary Outcome: MEN1309 Pharmacokinetic (PK) Parameter Vd
Description: volume of distribution based on the terminal phase
Time Frame: Cycle 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 3 | 4 | 1
L | 3.14 (0) | 6.69 (0) | 6.73 (0) | 49.47 (0) | 95.45 (0) | 4.97 (2.5) | 4.02 (1.32) | 4.73 (1.80) | 5.55 (3.24) | 5.08 (3.08) | 16.94 (0)

14. Other Pre Specified Outcome: Correlation of CD205 Expression in Tumors With Clinical Activity of MEN1309 Assessed According to RECIST 1.1 or Cheson Criteria (2014)
Description: Exploratory Endpoint: Correlation of CD205 expression in tumors with clinical activity of MEN1309 assessed according to RECIST 1.1 or Cheson Criteria (2014) in terms of Response Rate, Disease control rate, duration of response, overall survival, and progression free survival.
  N.B: No Data were available to assess this outcome.
Time Frame: Through study completion, from "August 28, 2017" to "January 8, 2020" (2 years and 4 months)
Population: N.B: No Data were available to assess this outcome.
Groups:
- STEP1 Solid Tumor All Doses + STEP 2 NHL: All Patients with CD205-positive advanced solid tumors inlcuded in STEP1 and all NHL patients included in STEP 2.
Arm/Group | STEP1 Solid Tumor All Doses + STEP 2 NHL
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Incidence of Anti-MEN1309 Antibodies
Description: Exploratory Endpoint: Immunogenicity analysis regarding the Incidence of anti-MEN1309 antibodies.
Time Frame: Day 1 of each Cycle (each cycle is 21 days)
Population: For this Outcome Results are not available per Cohorts, but only on the total of patients analyzed.
Measure: Number; unit: Patients
Arm/Group | STEP1 Solid Tumor All Doses + STEP 2 NHL
Number analyzed (Participants) | 28
Patients
  ADA Positive | 10
  ADA Negative | 18

ADVERSE EVENTS:
Time Frame: Through study completion, from "August 28, 2017" to "January 8, 2020" (2 years and 4 months)
Groups:
- Cohort1 0.05mg/kg STEP 1 Solid Tumors: Patients with CD205-advanced Solid Tumor, who recieved 0.05 mg/kg of MEN1309.
- Cohort2 0.10mg/kg STEP 1 Solid Tumors: Patients with CD205-advanced Solid Tumor, who recieved 0.10 mg/kg of MEN1309.
- Cohort3 0.20mg/kg STEP 1 Solid Tumors: Patients with CD205-advanced Solid Tumor, who recieved 0.20 mg/kg of MEN1309.
- Cohort4 0.40mg/kg STEP 1 Solid Tumors: Patients with CD205-advanced Solid Tumor, who recieved 0.40 mg/kg of MEN1309.
- Cohort5 0.80mg/kg STEP 1 Solid Tumors: Patients with CD205-advanced Solid Tumor, who recieved 0.80 mg/kg of MEN1309.
- Cohort6 1.60mg/kg STEP 1 Solid Tumors: Patients with CD205-advanced Solid Tumor, who recieved 1.60 mg/kg of MEN1309.
- Cohort7 2.40mg/kg STEP 1 Solid Tumors; Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF: Patients with CD205-advanced Solid Tumor, who recieved 2.40 mg/kg of MEN1309.
- Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF: Patients with CD205-advanced Solid Tumor, who recieved 3.36 mg/kg of MEN1309.
- Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF: Patients with CD205-advanced Solid Tumor, who recieved 2.00 mg/kg of MEN1309.
Arm/Group | Cohort1 0.05mg/kg STEP 1 Solid Tumors | Cohort2 0.10mg/kg STEP 1 Solid Tumors | Cohort3 0.20mg/kg STEP 1 Solid Tumors | Cohort4 0.40mg/kg STEP 1 Solid Tumors | Cohort5 0.80mg/kg STEP 1 Solid Tumors | Cohort6 1.60mg/kg STEP 1 Solid Tumors | Cohort7 2.40mg/kg STEP 1 Solid Tumors | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF | Cohort5 0.80mg/kg STEP 2 NHL
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/6 | 5/6 | 1/3 | 0/3 | 3/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1 | 1/1 | 0/1 | 5/6 | 5/6 | 3/3 | 3/3 | 2/4 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 1/1 | 1/1 | 6/6 | 6/6 | 3/3 | 3/3 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort1 0.05mg/kg STEP 1 Solid Tumors (N=1) | Cohort2 0.10mg/kg STEP 1 Solid Tumors (N=1) | Cohort3 0.20mg/kg STEP 1 Solid Tumors (N=1) | Cohort4 0.40mg/kg STEP 1 Solid Tumors (N=1) | Cohort5 0.80mg/kg STEP 1 Solid Tumors (N=1) | Cohort6 1.60mg/kg STEP 1 Solid Tumors (N=6) | Cohort7 2.40mg/kg STEP 1 Solid Tumors (N=6) | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF (N=3) | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF (N=3) | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF (N=4) | Cohort5 0.80mg/kg STEP 2 NHL (N=1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECOG performance Status Worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmunary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decrease appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort1 0.05mg/kg STEP 1 Solid Tumors (N=1) | Cohort2 0.10mg/kg STEP 1 Solid Tumors (N=1) | Cohort3 0.20mg/kg STEP 1 Solid Tumors (N=1) | Cohort4 0.40mg/kg STEP 1 Solid Tumors (N=1) | Cohort5 0.80mg/kg STEP 1 Solid Tumors (N=1) | Cohort6 1.60mg/kg STEP 1 Solid Tumors (N=6) | Cohort7 2.40mg/kg STEP 1 Solid Tumors (N=6) | Cohort8 3.36mg/kg STEP 1 Solid Tumors + GCSF (N=3) | Cohort7b 2.40mg/kg STEP 1 Solid Tumors +GCSF (N=3) | Cohort7c 2.00mg/kg STEP 1 Solid Tumors +GCSF (N=4) | Cohort5 0.80mg/kg STEP 2 NHL (N=1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Bliriubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
lymphocyte count decresed (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 6 (12) | 1 (1) | 1 (1) | 4 (7) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (3) | 1 (2)
white blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diorrhoea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Oedema Pheripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adnominal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesphageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT03403725/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03403725/SAP_001.pdf